CLINICAL TRIAL: NCT03177408
Title: Impact of HMGB1 on Diastolic Dysfunction in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jing Li (Other)
Responsible Party: Sponsor-Investigator, Jing Li, Doctor, Affiliated Hospital of Hebei University
Organization: Affiliated Hospital of Hebei University (Other)
Other Study IDs: 2017032901
Record Dates: First submitted 2017-04-16; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Diastolic Dysfunction; Hypertension; Inflammation
Keywords: Diastolic Dysfunction; Hypertension; HMGB1
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluated the association between HMGB1 and diastolic dysfunction in hypertensive patients. HMGB1 level were tested in all patients, and diastolic function determined by echocardiographic.

ELIGIBILITY:
Inclusion Criteria:

All of the hypertensive patients in both diastolic dysfunction and control groups were either newly diagnosed or were aware of hypertension without using any pharmacotherapy.

-

Exclusion Criteria:

Individuals already under treatment for hypertension were not include.

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample is recruited from the patients examined in the physical examination center of our hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences of HMGB1 levels between hypertensive patients with and without diastolic dysfunction | on the day of admission
  Blood samples of all individuals are collected on the day of admission and HMGB1 levels are tested. Echocardiographic assessment is performed with echocardiography device by using 2.5-3.5 Mega Hertz(MHz) transducer in the lateral decubitis position.

SECONDARY OUTCOMES:
Differences of HMGB1 levels between grades of diastolic dysfunction | on the day of admission
  Blood samples of all individuals are collected on the day of admission and HMGB1 levels are tested. Echocardiographic assessment is performed with echocardiography device by using 2.5-3.5 Mega Hertz(MHz) transducer in the lateral decubitis position.

IPD SHARING:
Plan to Share IPD: No